CLINICAL TRIAL: NCT02348268
Title: Myofascial Release Therapy in the Treatment of Occupational Mechanical Neck Pain: a Randomized Parallel Group Study.
Brief Title: Myofascial Release Therapy and Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FREMAP Mutual Insurance Company for Occupational Accidents and Diseases (Industry)
Collaborators: University of Vigo (Other); University Hospital A Coruña (Other)
Responsible Party: Principal Investigator, Iván Rodríguez Fuentes, Ph.D., FREMAP Mutual Insurance Company for Occupational Accidents and Diseases
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FREMAP
Record Dates: First submitted 2015-01-13; First posted 2015-01-28 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Neck Pain
Keywords: Neck Pain; Myofascial release; Manual therapy
MeSH Terms: conditions — Neck Pain | interventions — Musculoskeletal Manipulations; Myofascial Release Therapy; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual Therapy + Analgesic therapy (Active Comparator): The intervention for this group consisted of analgesic treatment in accordance with the guidelines of the FREMAP Protocol for the treatment of mechanical NP and additionally this group was treated with manual therapy (for 15 minutes).
  Interventions: Other: Manual Therapy; Device: Analgesic therapy
- Myofascial Release + Analgesic therapy (Experimental): The intervention for this group consisted of analgesic treatment in accordance with the guidelines of the FREMAP Protocol for the treatment of mechanical NP and additionally, this group was treated with myofascial release therapy (for 15 minutes).
  Interventions: Other: Myofascial Release Therapy; Device: Analgesic therapy

INTERVENTIONS:
Other: Manual Therapy — The manual therapy techniques included: (i) anterior-posterior and side-shift of the cervical spine; (ii) muscle energy technique involving side-bending of cervical spine; (iii) neuromuscular technique for restricted C1-C2 rotation; (iv) inhibitive occipital distraction; and (v) cervical stretching: post-isometric relaxation for the upper trapezius, scalene and sternocleidomastoid muscles.
  Arms: Manual Therapy + Analgesic therapy
Other: Myofascial Release Therapy — The myofascial release therapy techniques included: (i) cranial base release, adjusting the relation of the rectus capitis posterior muscles to the dura mater; (ii) gross release of the sternocleidomastoid muscle; (iii) release of the suprahyoid and infrahyoid muscles; and (iv) release of the retrohyoid fascia.
  Arms: Myofascial Release + Analgesic therapy
Device: Analgesic therapy — Analgesic therapy consisted of superficial thermotherapy by an infrared lamp (Infra 2000, Enraf Nonius) and TENS (TENSMED 911, Enraf Nonius). The 250-watts infrared lamp was focused at a distance of 50 cm on the cervical area for 15 minutes. TENS employed 80 Hz frequency, 150 µs pulse duration, with 50x50 mm electrodes (Gel-Trode, Enraf Nonius) placed on the painful or metamers areas for 20 minutes.
  Other Names: TENS + IRR

SUMMARY:
Mechanical neck pain is a musculoskeletal disorder usually associated with work absenteeism. Myofascial release therapy (MRT) is currently under development and has the treatment of mechanical neck pain as one of its main focal points. However, there is a paucity of studies reporting its effectiveness. For that purpose a randomized single-blind parallel group study was designed to compare the effectiveness of MRT with manual therapy (MT) for treating occupational mechanical neck pain. The sample (n=59) was randomly assigned to two therapeutic intervention programs. Group I patients were treated with MT and Group II patients were treated with MRT. Variables studied were intensity of neck pain, cervical disability, quality of life (QoL), craniovertebral angle and ranges of cervical motion.

DETAILED DESCRIPTION:
A variety of physiotherapy interventions have been used to treat mechanical neck pain (NP), but few of them have proven effective. The number of studies on the clinical effectiveness of MT techniques, such as myofascial release therapy (MRT), has seen a marked increase. MRT is a relatively new therapy with increasing acceptance and implementation in the daily clinical work of physiotherapists. However, there is a paucity of studies on biomechanical alterations associated with mechanical NP and its treatment with MRT, consequently, the clinical benefits of MRT remain unclear.

The purpose of this study was to assess the clinical efficacy of MRT in occupational mechanical NP and to determine if MRT has advantages over another MT protocol not including MRT.

An experimental parallel group study was designed. It was a single-blind (assessor) randomized controlled clinical trial. Patients from FREMAP - Mutual Insurance Company for Occupational Accidents and Diseases - participated in the study from January 2010 to December 2010. A total of 71 patients were asked to participate in the initial screening, but 8 did not meet inclusion criteria, 2 declined to participate in the study for personal reasons, and 2 could not participate for other reasons. 59 patients with NP were randomly distributed into two groups according to two therapeutic intervention programs. Group I (n=29; 18 females/11 males; mean age: 38.24 ± 11.35 years-old) was treated with MT and Group II (n=30; 15 females/15 males; mean age: 38.20 ± 10.70 years-old) was treated with MRT.

The intervention for both groups consisted of analgesic treatment in accordance with the guidelines of the FREMAP Protocol for the treatment of mechanical NP. The analgesic part of this protocol includes superficial thermotherapy (infrared lamp) and transcutaneous electrical stimulation (TENS). Additionally, Group I was treated with MT and Group II with MRT. There were 10 treatment sessions distributed within 4 successive weeks with three sessions being applied the first and third weeks and two sessions being applied the second and fourth weeks.

MT was provided by one physiotherapist, while MRT was performed by another physiotherapist, both from FREMAP. The sessions were held for nearly 50 minutes, until the completion of the intervention as determined by FREMAP.

Analgesic therapy consisted of the application of superficial thermotherapy by an infrared lamp (Infra 2000, Enraf Nonius) and TENS (TENSMED 911, Enraf Nonius). The 250-watts infrared lamp was focused at a distance of 50 cm on the cervical area for 15 minutes. TENS application employed 80 Hz frequency, 150 µs pulse duration, with 50x50 mm electrodes (Gel-Trode, Enraf Nonius) placed on the painful or metamers areas for 20 minutes.

The additional treatments were applied for both groups for 15 minutes. MT techniques included: (i) anterior-posterior and side-shift of the cervical spine; (ii) muscle energy technique involving side-bending of cervical spine; (iii) neuromuscular technique for restricted C1-C2 rotation; (iv) inhibitive occipital distraction; and (v) cervical stretching: post-isometric relaxation for the upper trapezius, scalene and sternocleidomastoid muscles.

The MRT included: (i) cranial base release, adjusting the relation of the rectus capitis posterior muscles to the dura mater (Hack et al., 1995); (ii) gross release of the sternocleidomastoid muscle; (iii) release of the suprahyoid and infrahyoid muscles; and (iv) release of the retrohyoid fascia.

ELIGIBILITY:
Inclusion Criteria:

* being between 18 and 65 years old; having mechanical neck pain with or without symptoms that radiated to the head and/or upper limbs (Guzman et al., 2009b); and
* scoring 10% or higher on the Neck Disability Index (NDI) or 2 points or more on the Visual Analogue Scale (VAS) of pain at initial evaluation (Farrar et al., 2001; Cleland et al., 2007).

Exclusion Criteria:

* Neck pain due to neoplasia, metastasis, severe osteoporosis, infectious or inflammatory processes, fractures, congenital anomalies, herniated disc, whiplash or cervical stenosis;
* evidence of cervical spinal cord compromise or radiculopathy; previous neck surgery;
* neck pain accompanied by dizziness caused by vertebrobasilar insufficiency or by headaches excluding those of cervical origin; and
* pregnant women. Patients were also excluded if they had received physiotherapy treatment in the previous three months; and had pending legal actions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Neck Pain | Baseline
  Assessed by the VAS, with a 2-point improvement being considered as clinically significant (Farrar et al., 2001; Cleland et al., 2007).

SECONDARY OUTCOMES:
Quality of life | Baseline
  Measured by the Short-Form Health Survey 36, (SF-36), which includes 8 dimensions: physical function (PF), role physical (RP), bodily pain (BP), general health (GH), mental health (MH), role emotional (RE), social functioning (SF) and vitality (VT), and comprises two global scales: the Physical Component Summary (PCS) and the Mental Component Summary (MCS) (Ware and Sherburne, 1992; Alonso et al., 1995; Hays et al., 1995).
Change from baseline Quality of life at 4 weeks | 4 weeks
  Measured by the Short-Form Health Survey 36, (SF-36), which includes 8 dimensions: physical function (PF), role physical (RP), bodily pain (BP), general health (GH), mental health (MH), role emotional (RE), social functioning (SF) and vitality (VT), and comprises two global scales: the Physical Component Summary (PCS) and the Mental Component Summary (MCS) (Ware and Sherburne, 1992; Alonso et al., 1995; Hays et al., 1995).
Cervical disability | Baseline
  Assessed by the Neck Disability Index (NDI), range of 0 to 50 and total scores expressed as a percentage (internal consistency of alfa: 0.74 to 0.93 and a minimum clinically difference of 5 points) (Westaway et al., 1998; Vernon, 2008).
Change from baseline cervical disability at 2 weeks | 2 weeks
  Assessed by the Neck Disability Index (NDI), range of 0 to 50 and total scores expressed as a percentage (internal consistency of alfa: 0.74 to 0.93 and a minimum clinically difference of 5 points) (Westaway et al., 1998; Vernon, 2008).
Change from baseline cervical disability at 4 weeks | 4 weeks
  Assessed by the Neck Disability Index (NDI), range of 0 to 50 and total scores expressed as a percentage (internal consistency of alfa: 0.74 to 0.93 and a minimum clinically difference of 5 points) (Westaway et al., 1998; Vernon, 2008).
Active cervical range of motion | Baseline
  Measured by a goniometer (SP-5060 CROM - cervical range of motion-, Performance Attainment Associates, St Paul, Minnesota, USA) (Haynes and Edmondston, 2002).
Change from baseline active cervical range of motion at 2 weeks | 2 weeks
  Measured by a goniometer (SP-5060 CROM - cervical range of motion-, Performance Attainment Associates, St Paul, Minnesota, USA) (Haynes and Edmondston, 2002).
Change from baseline active cervical range of motion at 4 weeks | 4 weeks
  Measured by a goniometer (SP-5060 CROM - cervical range of motion-, Performance Attainment Associates, St Paul, Minnesota, USA) (Haynes and Edmondston, 2002).
Craniovertebral angle | Baseline
  Assessed by a universal goniometer manufactured by 3B Scientific Products (Valencia, Spain) that incorporates a bubble level torpedo (Würth SA, Barcelona, Spain) (Wilmarth and Hilliard, 2002).
Change from baseline craniovertebral angle at 2 weeks | 2 weeks
  Assessed by a universal goniometer manufactured by 3B Scientific Products (Valencia, Spain) that incorporates a bubble level torpedo (Würth SA, Barcelona, Spain) (Wilmarth and Hilliard, 2002).
Change from baseline craniovertebral angle at 4 weeks | 4 weeks
  Assessed by a universal goniometer manufactured by 3B Scientific Products (Valencia, Spain) that incorporates a bubble level torpedo (Würth SA, Barcelona, Spain) (Wilmarth and Hilliard, 2002).
Change from baseline neck pain at 2 weeks. | 2 weeks
  Assessed by the VAS, with a 2-point improvement being considered as clinically significant (Farrar et al., 2001; Cleland et al., 2007).
Change from baseline neck pain at 4 weeks. | 4 weeks
  Assessed by the VAS, with a 2-point improvement being considered as clinically significant (Farrar et al., 2001; Cleland et al., 2007).

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J DeToro-Santos, Ph.D., Study Director — Department of Medicine, University of A Coruña.; Isaac M Fuentes-Boquete, Ph.D., Study Chair — Department of Medicine, University of A Coruña.; Iván Rodríguez-Fuentes, Ph.D., Principal Investigator — FREMAP Mutual Insurance Company for Occupational Accidents and Diseases
Locations (1):
- FREMAP - Mutual Insurance Company for Occupational Accidents and Diseases., A Coruña, A Coruña, Spain

REFERENCES:
- [Background] Lau HM, Wing Chiu TT, Lam TH. The effectiveness of thoracic manipulation on patients with chronic mechanical neck pain - a randomized controlled trial. Man Ther. 2011 Apr;16(2):141-7. doi: 10.1016/j.math.2010.08.003. Epub 2010 Sep 1. PMID 20813577
- [Background] Cleland JA, Glynn P, Whitman JM, Eberhart SL, MacDonald C, Childs JD. Short-term effects of thrust versus nonthrust mobilization/manipulation directed at the thoracic spine in patients with neck pain: a randomized clinical trial. Phys Ther. 2007 Apr;87(4):431-40. doi: 10.2522/ptj.20060217. Epub 2007 Mar 6. PMID 17341509
- [Background] Danto JB. Review of integrated neuromusculoskeletal release and the novel application of a segmental anterior/posterior approach in the thoracic, lumbar, and sacral regions. J Am Osteopath Assoc. 2003 Dec;103(12):583-96. PMID 14740981
- [Background] De-la-Llave-Rincon AI, Fernandez-de-las-Penas C, Palacios-Cena D, Cleland JA. Increased forward head posture and restricted cervical range of motion in patients with carpal tunnel syndrome. J Orthop Sports Phys Ther. 2009 Sep;39(9):658-64. doi: 10.2519/jospt.2009.3058. PMID 19721213
- [Background] Fernandez-de-las-Penas C, Hernandez-Barrera V, Alonso-Blanco C, Palacios-Cena D, Carrasco-Garrido P, Jimenez-Sanchez S, Jimenez-Garcia R. Prevalence of neck and low back pain in community-dwelling adults in Spain: a population-based national study. Spine (Phila Pa 1976). 2011 Feb 1;36(3):E213-9. doi: 10.1097/BRS.0b013e3181d952c2. PMID 21079541
- [Background] Gonzalez-Iglesias J, Fernandez-de-las-Penas C, Cleland JA, Alburquerque-Sendin F, Palomeque-del-Cerro L, Mendez-Sanchez R. Inclusion of thoracic spine thrust manipulation into an electro-therapy/thermal program for the management of patients with acute mechanical neck pain: a randomized clinical trial. Man Ther. 2009 Jun;14(3):306-13. doi: 10.1016/j.math.2008.04.006. Epub 2008 Aug 8. PMID 18692428
- [Background] Griegel-Morris P, Larson K, Mueller-Klaus K, Oatis CA. Incidence of common postural abnormalities in the cervical, shoulder, and thoracic regions and their association with pain in two age groups of healthy subjects. Phys Ther. 1992 Jun;72(6):425-31. doi: 10.1093/ptj/72.6.425. PMID 1589462
- [Background] Gross AR, Haines T, Goldsmith CH, Santaguida L, McLaughlin LM, Peloso P, Burnie S, Hoving J; Cervical Overview Group (COG). Knowledge to action: a challenge for neck pain treatment. J Orthop Sports Phys Ther. 2009 May;39(5):351-63. doi: 10.2519/jospt.2009.2831. PMID 19521013
- [Background] Gross A, Miller J, D'Sylva J, Burnie SJ, Goldsmith CH, Graham N, Haines T, Bronfort G, Hoving JL; COG. Manipulation or mobilisation for neck pain: a Cochrane Review. Man Ther. 2010 Aug;15(4):315-33. doi: 10.1016/j.math.2010.04.002. Epub 2010 May 26. PMID 20510644
- [Background] Guzman J, Haldeman S, Carroll LJ, Carragee EJ, Hurwitz EL, Peloso P, Nordin M, Cassidy JD, Holm LW, Cote P, van der Velde G, Hogg-Johnson S. Clinical practice implications of the Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders: from concepts and findings to recommendations. J Manipulative Physiol Ther. 2009 Feb;32(2 Suppl):S227-43. doi: 10.1016/j.jmpt.2008.11.023. PMID 19251069
- [Background] Hurwitz EL, Carragee EJ, van der Velde G, Carroll LJ, Nordin M, Guzman J, Peloso PM, Holm LW, Cote P, Hogg-Johnson S, Cassidy JD, Haldeman S. Treatment of neck pain: noninvasive interventions: results of the Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. J Manipulative Physiol Ther. 2009 Feb;32(2 Suppl):S141-75. doi: 10.1016/j.jmpt.2008.11.017. PMID 19251061
- [Background] Langevin HM, Cornbrooks CJ, Taatjes DJ. Fibroblasts form a body-wide cellular network. Histochem Cell Biol. 2004 Jul;122(1):7-15. doi: 10.1007/s00418-004-0667-z. Epub 2004 Jun 23. PMID 15221410
- [Background] Salt E, Wright C, Kelly S, Dean A. A systematic literature review on the effectiveness of non-invasive therapy for cervicobrachial pain. Man Ther. 2011 Feb;16(1):53-65. doi: 10.1016/j.math.2010.09.005. Epub 2010 Nov 12. PMID 21075037
- [Result] Ball TM. Structural integration-based fascial release efficacy in systemic lupus erythematosus (SLE): two case studies. J Bodyw Mov Ther. 2011 Apr;15(2):217-25. doi: 10.1016/j.jbmt.2010.10.006. Epub 2010 Nov 19. PMID 21419363
- [Result] Ercole B, Antonio S, Julie Ann D, Stecco C. How much time is required to modify a fascial fibrosis? J Bodyw Mov Ther. 2010 Oct;14(4):318-25. doi: 10.1016/j.jbmt.2010.04.006. Epub 2010 May 20. PMID 20850038
- [Result] Bronfort G, Evans R, Nelson B, Aker PD, Goldsmith CH, Vernon H. A randomized clinical trial of exercise and spinal manipulation for patients with chronic neck pain. Spine (Phila Pa 1976). 2001 Apr 1;26(7):788-97; discussion 798-9. doi: 10.1097/00007632-200104010-00020. PMID 11295901
- [Result] Castro-Sanchez AM, Mataran-Penarrocha GA, Granero-Molina J, Aguilera-Manrique G, Quesada-Rubio JM, Moreno-Lorenzo C. Benefits of massage-myofascial release therapy on pain, anxiety, quality of sleep, depression, and quality of life in patients with fibromyalgia. Evid Based Complement Alternat Med. 2011;2011:561753. doi: 10.1155/2011/561753. Epub 2010 Dec 28. PMID 21234327
- [Result] Day JA, Stecco C, Stecco A. Application of Fascial Manipulation technique in chronic shoulder pain--anatomical basis and clinical implications. J Bodyw Mov Ther. 2009 Apr;13(2):128-35. doi: 10.1016/j.jbmt.2008.04.044. Epub 2008 Jun 24. PMID 19329049
- [Result] Fernandez-de-las-Penas C, Alonso-Blanco C, Cuadrado ML, Pareja JA. Forward head posture and neck mobility in chronic tension-type headache: a blinded, controlled study. Cephalalgia. 2006 Mar;26(3):314-9. doi: 10.1111/j.1468-2982.2005.01042.x. PMID 16472338
- [Result] Fernandez-de-las-Penas C, Alonso-Blanco C, Cuadrado ML, Pareja JA. Neck mobility and forward head posture are not related to headache parameters in chronic tension-type headache. Cephalalgia. 2007 Feb;27(2):158-64. doi: 10.1111/j.1468-2982.2006.01247.x. PMID 17257237
- [Result] Fernandez-de-las-Penas C, Perez-de-Heredia M, Molero-Sanchez A, Miangolarra-Page JC. Performance of the craniocervical flexion test, forward head posture, and headache clinical parameters in patients with chronic tension-type headache: a pilot study. J Orthop Sports Phys Ther. 2007 Feb;37(2):33-9. doi: 10.2519/jospt.2007.2401. PMID 17366957
- [Result] Fletcher JP, Bandy WD. Intrarater reliability of CROM measurement of cervical spine active range of motion in persons with and without neck pain. J Orthop Sports Phys Ther. 2008 Oct;38(10):640-5. doi: 10.2519/jospt.2008.2680. PMID 18827326
- [Result] Gonzalez-Iglesias J, Fernandez-de-las-Penas C, Cleland JA, Gutierrez-Vega Mdel R. Thoracic spine manipulation for the management of patients with neck pain: a randomized clinical trial. J Orthop Sports Phys Ther. 2009 Jan;39(1):20-7. doi: 10.2519/jospt.2009.2914. PMID 19209478
- [Result] Hemmila HM. Bone setting for prolonged neck pain: a randomized clinical trial. J Manipulative Physiol Ther. 2005 Sep;28(7):508-15. doi: 10.1016/j.jmpt.2005.07.008. PMID 16182025
- [Result] Hoving JL, de Vet HC, Koes BW, Mameren Hv, Deville WL, van der Windt DA, Assendelft WJ, Pool JJ, Scholten RJ, Korthals-de Bos IB, Bouter LM. Manual therapy, physical therapy, or continued care by the general practitioner for patients with neck pain: long-term results from a pragmatic randomized clinical trial. Clin J Pain. 2006 May;22(4):370-7. doi: 10.1097/01.ajp.0000180185.79382.3f. PMID 16691091
- [Result] Lau KT, Cheung KY, Chan KB, Chan MH, Lo KY, Chiu TT. Relationships between sagittal postures of thoracic and cervical spine, presence of neck pain, neck pain severity and disability. Man Ther. 2010 Oct;15(5):457-62. doi: 10.1016/j.math.2010.03.009. PMID 20430685
- [Result] Leaver AM, Maher CG, Herbert RD, Latimer J, McAuley JH, Jull G, Refshauge KM. A randomized controlled trial comparing manipulation with mobilization for recent onset neck pain. Arch Phys Med Rehabil. 2010 Sep;91(9):1313-8. doi: 10.1016/j.apmr.2010.06.006. PMID 20801246
- [Result] Picelli A, Ledro G, Turrina A, Stecco C, Santilli V, Smania N. Effects of myofascial technique in patients with subacute whiplash associated disorders: a pilot study. Eur J Phys Rehabil Med. 2011 Dec;47(4):561-8. Epub 2011 Jul 28. PMID 21796089
- [Result] Ramos-Gonzalez E, Moreno-Lorenzo C, Mataran-Penarrocha GA, Guisado-Barrilao R, Aguilar-Ferrandiz ME, Castro-Sanchez AM. Comparative study on the effectiveness of myofascial release manual therapy and physical therapy for venous insufficiency in postmenopausal women. Complement Ther Med. 2012 Oct;20(5):291-8. doi: 10.1016/j.ctim.2012.03.005. Epub 2012 May 3. PMID 22863643
- [Result] Silva AG, Punt TD, Sharples P, Vilas-Boas JP, Johnson MI. Head posture and neck pain of chronic nontraumatic origin: a comparison between patients and pain-free persons. Arch Phys Med Rehabil. 2009 Apr;90(4):669-74. doi: 10.1016/j.apmr.2008.10.018. PMID 19345785
- [Result] Tozzi P, Bongiorno D, Vitturini C. Fascial release effects on patients with non-specific cervical or lumbar pain. J Bodyw Mov Ther. 2011 Oct;15(4):405-16. doi: 10.1016/j.jbmt.2010.11.003. Epub 2011 Jan 8. PMID 21943614
- [Result] Walker MJ, Boyles RE, Young BA, Strunce JB, Garber MB, Whitman JM, Deyle G, Wainner RS. The effectiveness of manual physical therapy and exercise for mechanical neck pain: a randomized clinical trial. Spine (Phila Pa 1976). 2008 Oct 15;33(22):2371-8. doi: 10.1097/BRS.0b013e318183391e. PMID 18923311
- [Result] Yip CH, Chiu TT, Poon AT. The relationship between head posture and severity and disability of patients with neck pain. Man Ther. 2008 May;13(2):148-54. doi: 10.1016/j.math.2006.11.002. Epub 2007 Mar 23. PMID 17368075
- [Derived] Rodriguez-Fuentes I, De Toro FJ, Rodriguez-Fuentes G, de Oliveira IM, Meijide-Failde R, Fuentes-Boquete IM. Myofascial Release Therapy in the Treatment of Occupational Mechanical Neck Pain: A Randomized Parallel Group Study. Am J Phys Med Rehabil. 2016 Jul;95(7):507-15. doi: 10.1097/PHM.0000000000000425. PMID 26745225